CLINICAL TRIAL: NCT06368141
Title: Neoadjuvant Chemotherapy Plus Sequential Immune Checkpoint Inhibitor (ICI) Therapy in Locally Advanced Colon Cancer
Acronym: NeoCHIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, PhD, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023294
Record Dates: First submitted 2023-11-27; First posted 2024-04-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoCHIC group (Experimental)
  Interventions: Drug: Serplulimab; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Serplulimab — Participants will receive a pre-operative CAPEOX and a sequential CAPEOX plus Serplulimab regimen.
  Other Names: HLX10
Drug: Capecitabine — Participants will receive a pre-operative CAPEOX and a sequential CAPEOX plus Serplulimab regimen.
Drug: Oxaliplatin — Participants will receive a pre-operative CAPEOX and a sequential CAPEOX plus Serplulimab regimen.

SUMMARY:
The goal of this clinical trial is to learn the effect of neoadjuvant chemotherapy plus sequential immune checkpoint inhibitor (ICI) therapy in locally advanced colon cancer. The main questions it aims to answer are:

* Does this neoadjuvant chemotherapy increase the pathologic complete response (pCR) of locally advanced colon cancer?
* Does this neoadjuvant chemotherapy improve the long-term survival of locally advanced colon cancer?

Participants will receive:

* a pre-operative CAPEOX (capecitabine oral + oxaliplatin i.v.)regimen.
* a sequential CAPEOX plus Serplulimab regimen.
* a standard complete mesocolic excision (CME) operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who volunteer to participate in this clinical trial and fully understand this study and sign the informed consent form (ICF), and willing to follow and capable of completing all testing procedures.
* Male or female aged 18-75 at the time of signing the ICF.
* Patients with histopathological confirmed primary colon adenocarcinoma
* MSS/RAS mutation patients with clinical stages T3N1-2 and T4N0-2
* an ECOG score of 0 or 1
* At least 1 measurable lesion according to RECIST 1.1 requirements.
* Patients must provide tumor tissue that meets the requirements for MSI/MMR testing.
* Expected survival period of at least 3 months.
* Negative hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) (-). If HBsAg (+) or HBcAb (+), hepatitis B virus deoxyribonucleic acid (HBV-DNA) must be <2500 copies/mL or 500 IU/mL before inclusion.
* Negative HCV antibody or HCV-RNA. If HCV-RNA is positive, the patient must have alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN to be included. Patients with co-infection of hepatitis B and hepatitis C should be excluded (HBsAg or HBcAb test is positive, and HCV antibody test is positive).
* Sufficient organ and bone marrow function confirmed by laboratory examinations within 7 days prior to the first use of the study medication, without severe hematopoietic abnormalities, heart, lung, liver, kidney dysfunction, and immune deficiency [no blood transfusion, albumin, recombinant human thrombopoietin, or colony stimulating factor (CSF) treatment was received within 14 days prior to the first use of the study medication]:

  1. Absolute value of neutrophils ≥ 1.5 × 109/L, platelet ≥ 100 × 109/L, hemoglobin concentration ≥ 9g/dL);
  2. Liver function test: bilirubin ≤ 1.5 × ULN; aspartate transaminase and glutamate transaminase ≤ 2.5 × ULN; if there is liver metastasis, AST and ALT ≤ 5 × ULN;
  3. Renal function test: serum creatinine ≤ 1.5 × ULN, or creatinine clearance rate (CCr) ≥ 60ml/min;
  4. Coagulation: international standardized ratio (INR) ≤ 1.5 × ULN, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
  5. Thyroid function: thyroid stimulating hormone (TSH) ≤ ULN; Should there be abnormalities, the levels of FT3 and FT4 should be examined. If the levels of FT3 and FT4 are normal, the patients can be included;
* Women of childbearing age must undergo a serum pregnancy test within 14 days before treatment, and the result is negative. And they are willing to use medically recognized effective contraceptive methods (such as intrauterine devices, contraceptives, or condoms) during the study period and within 3 months after the last dose of the study medication. For male subjects with partners of childbearing age, surgical sterilization is required, or it is recommended to use effective contraceptive methods during the study period and within 3 months after the last dose of the study medication.

Exclusion Criteria:

* Patients with recurrent colon cancer, or primary colon cancer who has received the following treatments before: radiation therapy for tumors, surgery, chemotherapy, immunotherapy or molecular targeted therapy, and other clinical research drugs
* Severe infection (such as conditions which require intravenous infusion of antibiotics, antifungal drugs, or antiviral drugs) within 4 weeks prior to treatment, or unexplained fever >38.5 ℃ during screening/initial administration;
* Hypertension without effective control through proper antihypertensive medication treatment (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg);
* Obvious clinical bleeding symptoms or obvious bleeding tendencies (bleeding>30 mL within 3 months, vomiting blood, black stool, bloody stool), hemoptysis (fresh blood>5 mL within 4 weeks), etc. within the first 3 months of treatment. Or patients with conditions that require long-term anticoagulant therapy with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day), such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep venous thrombosis, and pulmonary embolism.
* Active heart disease, including myocardial infarction and severe/unstable angina, occurred 6 months before treatment. Left ventricular ejection fraction<50% detected by echocardiography, with poor control of arrhythmia;
* Other malignant tumors within the past 5 years or at the same time (excluding cured skin basal cell carcinoma and cervical carcinoma in situ);
* Active or uncontrollable serious infections;
* Known human immunodeficiency virus (HIV) infection;
* Known clinically significant history of liver disease, including viral hepatitis [known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e. HBV DNA positivity (>1 × 104 copies/mL or>2000 IU/ml);
* Known hepatitis C virus infection (HCV) and HCV RNA positivity (>1 × 103 copies/mL), or other hepatitis or cirrhosis;
* III-IV cardiac insufficiency according to the New York Heart Association (NYHA) standard or left ventricular ejection fraction (LVEF)<50% according to color Doppler ultrasound examination;
* Patients with active pulmonary tuberculosis.
* Patients with past and current conditions such as interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, and severely impaired lung function that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
* The patient with known active or suspected autoimmune diseases. Patients with well controlled type I diabetes or immune related hypothyroidism who receive thyroid hormone replacement therapy are eligible. Patients with vitiligo who do not require intervention or with childhood asthma/allergies who have recovered without any intervention in adulthood are eligible.
* Patients who received live vaccine treatment within the first 28 days of enrollment.
* Patients who need to receive systemic corticosteroids (>10 mg/day prednisone efficacy dose) or other immunosuppressive drugs within the first 14 days of enrollment or during the study period.
* Any active infections that required systemic anti infective treatment, SARS-CoV-2 infection tested positive by RT-PCR within 14 days before the administration of the study drug. Subjects with a history of COVID-19 infection must have a negative RT-PCR test before the first administration of the study drug;
* History of major surgery within the first 28 days of randomization. The definition of major surgery in this study is that it requires at least 3 weeks of recovery time after surgery in order to receive surgery for treatment in this study.Patients who undergo tumor puncture or lymph node biopsy are eligible.
* Patient who has previously received treatment with other antibodies/drugs targeting immune checkpoints, such as PD-1, PD-L1, and cytotoxic T lymphocyte associated antigen 4 (CTLA-4).
* Patient who are currently participating in other clinical studies or planning to start treatment in this study less than 14 days from the end of the previous clinical study.
* Uncontrolled tumor related pain.
* History of severe allergies to any monoclonal antibody.
* History of allergies to any components of oxaliplatin and capecitabine.
* Women in pregnancy or lactating women.
* History of drug abuse of psychotropic substances or history of alcoholism.
* Any other disease with clinically significant metabolic abnormalities, physical examination abnormalities, or laboratory examination abnormalities, based on the judgment of the researcher, which is not suitable for the use of the study drug (such as having seizures and requiring treatment), or will affect the interpretation of the research results, or put the patient in a high-risk situation;
* Other factors that may cause the study to be terminated prematurely by the judgement of the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response | 2 weeks after operation
  pCR

CONTACTS AND LOCATIONS:
Overall Officials: Ren Zhao, PhD, Principal Investigator — Ruijin Hosipital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No